CLINICAL TRIAL: NCT02125669
Title: The Role of the 595 nm Pulsed Dye Laser in Treating Superficial Basal Cell Carcinomas at Low Risk Anatomical Sites: Outcome of a Double Blind Randomized Placebo Controlled Trial
Brief Title: Pulsed Dye Laser in Treating Superficial Basal Cell Carcinomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hautklinik Darmstadt (Other)
Collaborators: University Medicine Greifswald (Other)
Responsible Party: Principal Investigator, Maurizio Podda, PD Dr. med., Hautklinik Darmstadt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FF57/2012
Record Dates: First submitted 2014-04-13; First posted 2014-04-29 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Basal Cell Carcinoma
Keywords: basal cell carcinoma; laser surgery; pulsed dye laser; randomized controlled trial
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laser Treatment (Active Comparator): Pulsed dye laser 595nm
  Interventions: Procedure: Laser treatment
- SHAM Treatment (Sham Comparator): using the pulsed dye laser (PDL) laser without releasing a pulse
  Interventions: Device: SHAM-Treatment

INTERVENTIONS:
Procedure: Laser treatment — Pulsed dye laser 595nm
  Arms: Laser Treatment
Device: SHAM-Treatment — using the pulsed dye laser (PDL) laser without releasing a pulse
  Arms: SHAM Treatment

SUMMARY:
Pulsed dye laser (PDL) treatments have been suggested to be a safe and effective therapeutic approach for treating basal cell carcinomas. Robust supporting evidence is, however, lacking due to inconsistent design of available studies. The purpose of this study is to evaluate the PDL's efficacy and safety in treating superficial basal cell carcinoma (sBCC) at low risk anatomical sites in an evidence based study setting.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed unpigmented sBCC on the trunk and extremities
* maximal tumour diameter 30 mm

Exclusion Criteria:

* Fitzpatrick skin type >III
* pregnancy
* previous BCC treatment within 4 weeks
* coagulation disorders
* photo sensitizing medication
* any indication of poor compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
complete response | 9 months

SECONDARY OUTCOMES:
patients satisfaction | 9 months
  questionnaire
side effects | 9 months
  questionnaire
reduction of tumor diameter and tumor thickness | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Podda, Dr., Principal Investigator — Hautklinik Darmstadt; Syrus Karsai, Dr., Study Director — Hautklinik Darmstadt; Heiko Friedl, Study Chair — Hautklinik Darmstadt